CLINICAL TRIAL: NCT06908382
Title: A Single-Arm Study of Iparomlimab and Tuvonralimab (QL1706) in Combination With Chemotherapy as Neoadjuvant Therapy for Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant QL1706 Therapy for ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Yang Zhe, Tumor Research and Therapy Center, Shandong Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWYX-20241055
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Resectable Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection — QL1706 (5 mg/kg, q3w) +Paclitaxel for injection (albumin bound) (260mg/m2 D1, q3w)+cisplatin (75mg/m2 D1, q3w)/carboplatin (AUC 5 D1) ， 3 cycles

SUMMARY:
This study plans to enroll 32 patients with resectable esophageal squamous cell carcinoma. The treatment regimen consists of Iparomlimab and Tuvonralimab(QL1706) combined with chemotherapy: intravenous infusion of QL1706 (5 mg/kg, q3w) in combination with albumin-bound paclitaxel (260 mg/m² on day 1, q3w) plus cisplatin (75 mg/m² on day 1, q3w) or carboplatin (AUC 5 on day 1, q3w) for 3 cycles. Surgical resection will be performed 3-6 weeks after treatment completion. Pre-treatment and surgical tissue specimens will be collected for analysis of tumor immune microenvironment changes using digital gene quantification technology. Peripheral blood samples will be obtained for dynamic ctDNA monitoring at four time points: within 7 days pre-treatment, 7 days pre-surgery, 7-30 days post-surgery, and 6 months post-surgery. The primary endpoint is the pathological complete response (pCR) rate, and secondary endpoints include major pathological response (MPR) and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form to voluntarily join this study;
2. Age 18-75 years old, male or female;
3. ECOG PS 0-1;
4. Planned surgical treatment after completion of neoadjuvant therapy;
5. Patients with esophageal squamous cell carcinoma diagnosed pathologically as ct1b-ct2n+or ct3-ct4a any nm0

Exclusion Criteria:

1. The subject has any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; the subject suffers from vitiligo; asthma has been completely relieved in childhood and does not need any intervention after adulthood can be included, but asthma that needs bronchodilators for medical intervention cannot be included);
2. The subjects are using immunosuppressive agents or systemic or absorbable local hormones to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other effective hormones), and continue to use them within 2 weeks before enrollment;
3. Severe allergic reaction to other monoclonal antibodies;
4. There are cardiac clinical symptoms or diseases that are not well controlled, such as: (1) heart failure above NYHA grade 2 (2) unstable angina pectoris (3) myocardial infarction within one year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention (5) qtc>450ms (male); Qtc>470ms (female);
5. Patients at risk of massive bleeding
6. Abnormal coagulation function (inr>1.5 or pt>16s), bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
7. Genetic or known to exist Acquired hemorrhage and thrombotic tendency (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.) or arteriovenous thrombosis events in recent 6 months (until the first use of shr-1210);
8. Subjects with active infection or fever of unknown origin>38.5 degrees during screening and before the first administration;
9. Patients with previous and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe impairment of lung function;
10. Subjects with congenital or acquired immune deficiency (such as HIV infected), or active hepatitis (hepatitis B reference: HBV DNA detection value exceeds the upper limit of normal value; Hepatitis C reference: HCV virus titer or RNA detection value exceeds the upper limit of normal value);
11. Those who have used other drugs in clinical trials within 4 weeks before the first medication;
12. The subjects had previously or simultaneously suffered from other malignant tumors;
13. Subjects may receive other systemic anti-tumor treatment during the study period;
14. The subjects had previously received other PD-1 antibody therapy or other immunotherapy for PD-1/PD-L1;
15. Live vaccines were administered less than 4 weeks before the study or during the study period;
16. According to the judgment of the investigator, the subject has other factors that may lead to the forced termination of this study, such as other serious diseases (including mental diseases) requiring combined treatment, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR Rate | one month after esophageal cancer surgery
  The rate of patients with primary tumor and lymph nodes both achieved pathological complete response

SECONDARY OUTCOMES:
MPR Rate | one month after esophageal cancer surgery
  The percentage of subjects with less than 10% tumor residue in the primary tumor site
EFS | approximately 5 years
  The time from initial drug use to the occurrence of events as defined by the study protocol
OS | approximately 6 years
  The time from initial drug use to death due to any cause
Safety (adverse event) | From initial drug use to one month after surgery
  Rate of adverse event and severe event according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No